CLINICAL TRIAL: NCT00772616
Title: Influence of Intraoperative Analgesia (Sufentanil Administered According to the Usual Criteria or Remifentanil Administered by a Closed-loop System Using Bispectral Index as the Controller) on the Postoperative Morphine Consumption
Brief Title: Influence of Intraoperative Analgesia on the Postoperative Morphine Consumption
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2007/13
Record Dates: First submitted 2008-10-11; First posted 2008-10-15 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia
Keywords: Anesthesia; Analgesia; Patient-Controlled Analgesia; Hyperalgesia
MeSH Terms: conditions — Agnosia; Hyperalgesia | interventions — Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients will receive propofol and remifentanil automatically administered (closed-loop administration using bispectral index as the single input for the controller).
  Interventions: Drug: Remifentanil
- 2 (Active Comparator): Patients will receive propofol automatically administered (closed-loop administration using bispectral index as the single input for the controller) and sufentanil according to usual criteria
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Remifentanil — closed-loop administration using bispectral index as the single input for the controller.
  Arms: 1
Drug: Sufentanil — dosage according to usual criteria
  Arms: 2

SUMMARY:
Unlike longer acting opiates (sufentanil), remifentanil may provoke postoperative hyperalgesia. We have developed two automated bispectral index - guided drug delivery systems: one for propofol administration, the other for combined propofol and remifentanil administration. Both systems achieve the same objective: similar level of anesthesia indicated by bispectral index levels between 40 to 60. We make the assumption that this method of automated remifentanil administration may avoid postoperative hyperalgesia. Patients scheduled for abdominal surgery will be divided into two groups:

* in one group, patients will receive automatically delivered propofol and manually delivered sufentanil according to the usual criteria,
* in the other group, patients will receive propofol and remifentanil both automatically administered.

Assessment of postoperative hyperalgesia will be primarily based on morphine consumption (patient controlled analgesia) and detection of cutaneous hyperalgesia areas.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for an abdominal surgery

Exclusion Criteria:

* Age less than 18 years,
* Pregnant women,
* Allergy to propofol, sufentanil, remifentanil, morphine, muscle relaxant, or to a component,
* Hypersensibility to sufentanil, remifentanil or to a derivate of fentanyl,
* Inflammatory bowel disease,
* Chronic pain,
* Patients receiving a psychotropic treatment or a a morphine agonist-antagonist,
* Alcoholic patients and patients taking opiates,
* History of neurological disorders or central brain lesion, of severe respiratory insufficiency, of hepatic insufficiency,
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Dose of morphine administered during the postoperative period (patient controlled analgesia) | 48 postoperative hours

SECONDARY OUTCOMES:
postoperative pain scores | 48 postoperative hours
postoperative hyperalgesia | up to 5th to 7th postoperative days
nausea vomiting | 48 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

REFERENCES:
- [Background] Joly V, Richebe P, Guignard B, Fletcher D, Maurette P, Sessler DI, Chauvin M. Remifentanil-induced postoperative hyperalgesia and its prevention with small-dose ketamine. Anesthesiology. 2005 Jul;103(1):147-55. doi: 10.1097/00000542-200507000-00022. PMID 15983467
- [Background] Liu N, Chazot T, Genty A, Landais A, Restoux A, McGee K, Laloe PA, Trillat B, Barvais L, Fischler M. Titration of propofol for anesthetic induction and maintenance guided by the bispectral index: closed-loop versus manual control: a prospective, randomized, multicenter study. Anesthesiology. 2006 Apr;104(4):686-95. doi: 10.1097/00000542-200604000-00012. PMID 16571963